CLINICAL TRIAL: NCT04521088
Title: Epidemiological Analysis of Ambulant Patients in a COVID-19 Outpatient Clinic
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Principal Investigator, Prof. Randerath, Prof. Dr., Wissenschaftliches Institut Bethanien e.V
Other Study IDs: WI-1252
Record Dates: First submitted 2020-07-02; First posted 2020-08-20 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- visitors of the outpatient clinic for COVID-19: visitors of the outpatient clinic for COVID-19

SUMMARY:
There is insufficient knowledge about transmission routes and the effectiveness of general protective measures to prevent infection, such as the closure of schools or the wearing of mouthguards. This will be illustrated using the example of the COVID-19 outpatient clinic in Solingen and the positive COVID-19 tests registered there.

Another aspect we would like to address in this study is the number of COVID-19 tests performed against the background of political events or dramatic accumulations of COVID-19 cases in other parts of Germany or Europe. Do speeches by political leaders about the COVID-19 situation or a very strong regional spread of infection elsewhere have an impact on the frequency with which people react sensitively to suspicious symptoms and undergo testing for infection?

DETAILED DESCRIPTION:
The aim of this study is to analyse the frequency of positive COVID-19 tests and the infection chains in Solingen since February 2020:

1. a prospective survey (telephone contact) of the positively tested patients is done to analyze the social environment and thus provide information about possible transmission routes. Is transmission mainly within the family through visits from relatives or rather through large extra-familial gatherings, such as in the case of the open huts and après-ski bars in Ischgl? Are there age- or gender-specific transmission routes (personal habits, travel)?
2. analysis of the number of positive tests in connection with general measures to contain the infection (closure of schools, mouthguards obligation, etc.)
3. characterization of positively tested patients based on anthropometric data and medical history.
4. the effect of political events and developments in world affairs on the daily visitor frequency in the COVID-19 outpatient clinic will be retrospectively investigated. Is there an accumulation of tests after speeches by politicians or public figures (Angela Merkel, Armin Laschet, Queen Elizabeth II, etc.) or after dramatic infection numbers in other parts of Germany or Europe (Heinsberg, Ischgl, etc.)?

ELIGIBILITY:
Inclusion Criteria:

* positive COVID-19 test result

Exclusion Criteria:

* negative COVID-19 test result
* Any medical, psychological or other condition which restricts the ability to provide information or consent of the patient for voluntary participation in this examination

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all visitors of the outpatient clinic for COVID-19 since february 2020 in Solingen
Sampling Method: Non-Probability Sample
Enrollment: 1316 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
possible risk factors | 0-4 weeks
  medical history and medication of positive tested patients
frequency of positive test results after prescribed protective measures | about 8 months
  frequency of positive test results after prescribed protective measures
frequency of positive test results within the family or other social groups | about 8 months
  frequency of positive test results within the family or other social groups

SECONDARY OUTCOMES:
number of COVID-19 tests in the outpatient clinic | about 8 months
  number of COVID-19 tests in the outpatient clinic against the background of events in world affairs

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Pneumologie an der Universität zu Köln / Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No